CLINICAL TRIAL: NCT00886730
Title: Feasibility Study of Methods of Referral Primary Care Patients With Depression for Internet-Based Social Support
Brief Title: Primary Care Patients With Depression for Internet-Based Social Support
Acronym: Psychobabble
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15836A; R34MH073742-01 (NIH)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Depressive Disorder
Keywords: Depressive disorder; Primary care; Internet; Social support; Feasibility
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Simple Card (Experimental): Participants will receive a simple 3"x5" card with the name of the website and the following description. "www.psychobabble.com (or new name). A website to help individuals with depression recover."
  Interventions: Behavioral: Simple Card
- Patient Centered Brochure (Experimental): Participants will receive an 8"x11" handout that provides a more complete description of the depression website. The handout will be based on a patient perspective with samples of Internet postings from users. This card will emphasize peer-to-peer support and not mention health care organizations or health care provider endorsements. The information will address potential barriers to use: user will not be identified, posting will not take that much time, information from peers can be checked for accuracy with other peers and providers, and helping patient learn how to tell their usual health care providers about their activities on the Internet site. Participants will be asked to provide their email so a reminder about the Internet depression site can be emailed to them at 1 week and 2 weeks. They will still be part of the study even if they will not provide their email.
  Interventions: Behavioral: Patient Centered Brochure
- Physicians endorsement (Experimental): Participants will include the same card in experimental group 2 with the addition of a personal endorsement by the patient's health care provider in the form of a standardized letter signed by the physician. Participants will be asked to provide their email so a reminder about the Internet depression site can be emailed to them at 1 week and 2 weeks.
  Interventions: Behavioral: Physician's endorsement

INTERVENTIONS:
Behavioral: Simple Card — Participants will receive a simple 3"x5" card with the name of the website and the following description. "www.psychobabble.com (or new name). A website to help individuals with depression recover."
  Arms: Simple Card
Behavioral: Patient Centered Brochure — Participants will receive an 8"x11" handout that provides a more complete description of the depression website. The handout will be based on a patient perspective with samples of Internet postings from users. This card will emphasize peer-to-peer support and not mention health care organizations or health care provider endorsements. The information will address potential barriers to use: user will not be identified, posting will not take that much time, information from peers can be checked for accuracy with other peers and providers, and helping patient learn how to tell their usual health care providers about their activities on the Internet site. Participants will be asked to provide their email so a reminder about the Internet depression site can be emailed to them at 1 week and 2 weeks. They will still be part of the study even if they will not provide their email.
  Arms: Patient Centered Brochure
Behavioral: Physician's endorsement — Participants will include the same card in experimental group 2 with the addition of a personal endorsement by the patient's health care provider in the form of a standardized letter signed by the physician. Participants will be asked to provide their email so a reminder about the Internet depression site can be emailed to them at 1 week and 2 weeks.
  Arms: Physicians endorsement

SUMMARY:
The purpose of this study is to develop and pilot test two interventions that lead to at least 30% of individuals with depression presenting to primary care engaging with an Internet-based depression support group. The investigators will identify primary care patients with depression who state they have access to the Internet and are willing to consider treatment for depression. In the primary care office they will be given one of three interventions introducing them to the Internet depression support group site. The major outcome will be accessing the depression Internet support group at least once in the following four weeks.

The results of this study will provide important information on whether it is possible to recruit a substantial proportion of primary care patients to engage in a potentially useful and inexpensive addition to standard depression care. If this is not possible, the likelihood of successfully completing a RCT of the effectiveness of depression Internet support groups utilizing primary care patients would be low. Researchers trying to assess the effectiveness of depression Internet support groups would have to go to alternative designs such as recruiting patients with depression as they try to join the depression Internet support groups and randomizing some to a delay in joining the group.

DETAILED DESCRIPTION:
Our specific aim is to develop and pilot test two interventions that lead to at least 30% of individuals with depression presenting to primary care engaging with an Internet-based depression support group. We will identify primary care patients with depression who state they have access to the Internet and are willing to consider treatment or are currently in treatment for depression. In the primary care office they will be given one of three interventions introducing them to the Internet depression support group site. Patients will be randomized to three experimental groups: 1) simple card with only the name of the web address; 2) 8"x11" paper with screen shots of the Internet site home page, a list of features provided by the site, and two patient stories describing how the Internet site helped them; and 3) the 8"x11" announcement (from intervention 2) plus endorsement of the site by the primary care provider. The last two interventions will also ask patients to provide an email address so one email reminder can be sent to them. The major outcome will be accessing the depression Internet support group at least once in the following four weeks.

The results of this study will provide important information on whether it is possible to recruit a substantial proportion of primary care patients to engage in a potentially useful and inexpensive addition to standard depression care. If this is not possible, the likelihood of successfully completing a RCT of the effectiveness of depression Internet support groups utilizing primary care patients would be low. Researchers trying to assess the effectiveness of depression Internet support groups would have to go to alternative designs such as recruiting patients with depression as they try to join the depression Internet support groups and randomizing some to a delay in joining the group. We will also use this study to learn more about what patient characteristics are associated with engaging with an internet depression support group. While the focus of this study is Psychobabble, the intent of the study is to explore ease of referral, predictors of use and participant experiences as may relate to the general concept of Internet-based social support.

Specific AIM 1: We believe that participants randomized to the either that 8 x 11" brochure or the recommendation by the primary care physician will be more likely to visit and use the site than those who receive only a recommendation card (50% versus 35% versus 10%). We hypothesize that greater levels of encouragement/recommendation will be associated with higher levels of internet site usage. A sample size of 225 (N-110 at University of Chicago and N=115 at Johns Hopkins) will have power of 0.8 to detect the difference between either the card group or the brochure or physician recommendation group.

Specific Aim 2: We believe that those with higher self-efficacy and greater levels of trust in their primary care physician will be more likely to visit the site one time. We will conduct a logistic regression analysis to determine whether base self-efficacy and greater levels of trust predict use of the internet site after adjusting for group assignment. We hypothesize that higher levels of self-efficacy and physician trust will be associated with greater internet site use. Will believe a total N=225 will be sufficient to evaluate the relationship between 10 independent variables and the outcome of site usage (<15 cells/variable).

Specific Aim 3: We will determine if an internet based social support group is acceptable and feasible for primary care patients. Specifically, we will evaluate whether the internet site increased their knowledge of, or motivation for, depression treatment (Change in level of agreement to with regard to "accepting my doctors diagnosis of depression", strongly disagree 1, strongly agree 5). We hypothesize that levels of agreement will increase pre to post-study. A sample size of 225 (N=110 at University of Chicago and N=115 at Johns Hopkins) will have power of 0.8 to detect the difference of agree (4) pre-study to (5) strongly agree post study.

Specific Aim 4: We believe that social support and knowledge gained on the internet may influence subsequent care seeking or coping behaviors. Specifically, we will evaluate whether they have sought care or adopted coping skills 6 weeks after study entry. We hypothesize that both these behaviors will increase from pre to post study. A sample size of 225 (N=110 at University of Chicago and N=115 at Johns Hopkins) will have power of 0.8 to detect the difference of treatment participation pre-study of 0.4 versus 0.65 post study.

Specific Aim 5: We believe that social support or knowledge gained on the internet site leading to changed behaviors may results in lower levels of depressed mood. Specifically, we will compare levels of depressed mood at baseline and at 6 week follow-up. We hypothesize that their will be modest decline in depressed mood from pre study baseline to post study. A sample size of 225 (N=110 at University of Chicago and N=115 at Johns Hopkins) will have power of 0.8 to detect the difference of treatment participation pre study CES-D score of 24 post study score of 20.

ELIGIBILITY:
Inclusion Criteria:

1. PHQ score of 8 or above with either depressed mood or anhedonia/and or is considering treatment for depressed mood,
2. does not reject all treatment for depression,
3. has not viewed or posted messages more than once in the last month on any Internet depression support group website,
4. does not self-report diagnoses of bipolar disorder by a health professional,
5. age 18 years or older,
6. attends a primary care clinic and have visited in last 6 months, AND
7. has Internet access for the next four weeks, has been on the Internet at least three times, and has used email by him/herself. We are slightly lowering the PHQ score from the usual 10 (cutoff for major depression) to 8 because we know treatment for depression is frequently initiated for those who do not meet formal criteria for major depression. However we are only including patients with PHQ scores below the usual cutoff for major depression if they are currently receiving or are considering some form of depression treatment. University of Chicago students will need to identify their primary care provider to be enrolled in the study.

Exclusion Criteria:

1. active bipolar disorder,
2. those with no access to the internet,
3. those who state they are not under treatment nor would they consider any form of treatment, OR
4. those considered to be at high risk of suicide attempts. These include those with past psychiatric hospitalization, past suicide attempts, bipolar disorder or score of greater than 1 on the PHQ-9 suicide assessment or who reports intent for self-harm as per assessment in the suicide prevention protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Percentage visiting the Internet site | 6 weeks

SECONDARY OUTCOMES:
Feasibility, helpfulness and safety of Internet site | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Physician's Group - PCG Maryland Avenue, Chicago, Illinois, United States

REFERENCES:
- [Derived] Van Voorhees BW, Hsiung RC, Marko-Holguin M, Houston TK, Fogel J, Lee R, Ford DE. Internal versus external motivation in referral of primary care patients with depression to an internet support group: randomized controlled trial. J Med Internet Res. 2013 Mar 12;15(3):e42. doi: 10.2196/jmir.2197. PMID 23482332